CLINICAL TRIAL: NCT06778187
Title: A Phase 2 Study of Oral Arsenic Trioxide (Arsenol ®)-Based Low-intensity Treatment for Previously Untreated or Relapsed/Refractory TP53-mutated Myeloid Malignancies
Brief Title: Oral-ATO for TP53-mutated Myeloid Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATO-IIS001
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Neoplasm; Chronic Myelomonocytic Leukemia; TP53 Gene Mutation; Arsenic Trioxide
Keywords: Acute myeloid leukemia; Myelodysplastic neoplasm; Chronic myelomonocytic leukemia; TP53 mutation; Oral arsenic trioxide
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral arsenic trixoide (Experimental): Patients will be treated in 28-day cycles.
  Each cycles will comprise:
  Oral ATO (10mg/day or 0.15mg/kg/day in patients < 50kg) from Days 1-14
  PLUS:
  * Oral ascorbic acid (1000mg/day) from Days 1-14
  * Azacitidine (75mg/m2/day s.c. or i.v.) from days 1-7; OR Decitabine (20mg/m2/day i.v.) from days 1-5; OR Oral-decitabine-cedazuridine (1 tablet/day) from days 1-5.
  * Venetoclax (100mg-400mg/day) from Days 1-14 (if used)
  Interventions: Drug: Oral arsenic trioxide

INTERVENTIONS:
Drug: Oral arsenic trioxide — Patients will be treated in 28-day cycles.
  Each cycles will comprise:
  Oral arsenic trixoide (10mg/day or 0.15mg/kg/day in patients < 50kg) from Days 1-14
  PLUS:
  * Oral ascorbic acid (1000mg/day) from Days 1-14
  * Azacitidine (75mg/m2/day s.c. or i.v.) from days 1-7; OR Decitabine (20mg/m2/day i.v.) from days 1-5; OR Oral-decitabine-cedazuridine (1 tablet/day) from days 1-5.
  * Venetoclax (100mg-400mg/day) from Days 1-14 (if used)

SUMMARY:
This is an open-label, phase 2 study of oral arsenic trioxide (Arsenol ®) in combination with ascorbic acid and investigator choice of low-intensity therapy in patients with previously untreated or relapse/refractory TP53-mutated acute myeloid leukemia (AML), myelodysplastic neoplasm (MDS), chronic myelomonocytic leukemia (CMML).

DETAILED DESCRIPTION:
Approximately 30 patients will be enrolled prospectively. Approximately 15 patients will be previously untreated and 15 patients will be relapsed or refractory to 1 or more lines of therapy.

Oral arsenic trioxide (oral-ATO) (Arsenol ®) will be used in combination with ascorbic acid, and investigator choice of low-intensity therapy that comprised hypomethylating agent (HMA) with or without venetoclax. The choice of hypomethylating agents include subcutaneous (s.c.) / intravenous (i.v.) azacitidine, i.v. decitabine or oral-decitabine-cedazuridine. Patients will be treated in 28-day days cycles.

Pending study team review of the tolerability, hematologic response, and molecular response to the combination, a future randomized Phase 2 efficacy study may be planned.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Age ≥18 years
3. Diagnosis of acute myeloid leukemia (AML), myelodysplastic neoplasm (MDS) or chronic myelonocytic leukaemia (CMML) by World Health Organization (WHO) 2022 criteria (1, 3)
4. Presence of TP53 mutation
5. Previously untreated patients for Cohort A (Treatment-naïve), or Patients failing 1 or more lines of prior treatment for Cohort B (Relapsed and Refractory)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Women of childbearing potential and fertile men must agree to use an approved method of contraception from Screening until 30 days after the last dose of oral arsenic trioxide, ascorbic acid, venetoclax and azacitidine/decitabine/oral-decitabine-cedazuridine.

Exclusion Criteria:

Inclusion Criteria

1. Willing and able to provide informed consent
2. Age ≥18 years
3. Diagnosis of acute myeloid leukemia (AML), myelodysplastic neoplasm (MDS) or chronic myelonocytic leukaemia (CMML) by World Health Organization (WHO) 2022 criteria (1, 3)
4. Presence of TP53 mutation
5. Previously untreated patients for Cohort A (Treatment-naïve), or Patients failing 1 or more lines of prior treatment for Cohort B (Relapsed and Refractory)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
7. Women of childbearing potential and fertile men must agree to use an approved method of contraception from Screening until 30 days after the last dose of oral arsenic trioxide, ascorbic acid, venetoclax and azacitidine/decitabine/oral-decitabine-cedazuridine.

Exclusion Criteria

1. Use of an investigational agent within 14 days of study treatment (or at least 7 half-lives of that agent, whichever is longer), prior to the first dose of oral arsenic trioxide
2. Known hypersensitivity to arsenic trioxide, ascorbic acid, venetoclax or azacitidine/decitabine/oral-decitabine-cedazuridine or their excipients.
3. Uncontrolled, active infection
4. Major surgery within 4 weeks of starting the study drug, or not recovered from side effects of surgery
5. Any other serious medical conditions that could compromise study participation, in the opinion of the investigator
6. Known HIV infection or known, active hepatitis B or hepatitis C infection
7. Concurrent second active and non-stable malignancy (patients with a concurrent second active but stable malignancy, i.e., non-melanoma skin cancers, are eligible)
8. Known history of long QT syndrome (LQTS) or corrected QT interval by Fridericia formula (QTcF) ≥ 480 ms
9. Evidence at the time of Screening of significant renal or hepatic insufficiency (unless due to hemolysis) as defined by any of the following local laboratory parameters:

   1. Calculated glomerular filtration rate (GFR; using the Cockcroft-Gault equation or eGFR; using CKD-EPI) < 40 mL/min
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 x the local upper limit of normal
10. Pregnant or lactating females, or females planning to become pregnant at any time during the study
11. Unwilling or unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 24 months
  Enumeration and description of adverse events (AEs), serious adverse events (SAEs), and other AEs

SECONDARY OUTCOMES:
Response rates | 24 months
  Proportion of patients who achieve a response by European LeukemiaNet (ELN) criteria (for AML) and International Working Group (IWG) criteria (for MDS and CMML)
Rates of molecular responses | 24 months
  Changes in mutant allele frequencies of TP53 mutations and other co-mutations during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Gill, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality issues.

REFERENCES:
- [Background] Sallman DA, Stahl M. TP53-mutated acute myeloid leukemia: how can we improve outcomes? Blood. 2025 Jun 12;145(24):2828-2833. doi: 10.1182/blood.2024024245. PMID 39236289